CLINICAL TRIAL: NCT03884881
Title: The Role of Second-generation Sequencing in the Treatment of Severe Pneumonia With Initial Treatment Failure
Brief Title: Second-generation Sequencing Guides the Treatment of Severe Pneumonia
Acronym: NGS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 81770080
Record Dates: First submitted 2019-03-14; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2018-12

CONDITIONS: Pneumonia; Metagenomic Next Generation Sequencing
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- metagenomic next generation sequencing (Other): Adjust medication for patients with severe pneumonia based on mNGS results
  Interventions: Diagnostic Test: metagenomic next generation sequencing; Drug: Meropenem，Imipenem，Caspofene，Osstat
- Conventional pathogen detection (Other): Blood, bronchoalveolar lavage fluid (BALF), bronchial secretions samples will be collected and microbiologically tested prior to initial empirical antibiotic use.
  Interventions: Diagnostic Test: Conventional pathogen detection; Drug: Meropenem，Imipenem，Caspofene，Osstat

INTERVENTIONS:
Diagnostic Test: metagenomic next generation sequencing — Pathogens in the NGS group will be tested by NGS，then according the NGS results, adjust antibiotics
  Arms: metagenomic next generation sequencing
Diagnostic Test: Conventional pathogen detection — Morphological detection, microbial culture, nucleic acid amplification technology, serological pathogen antibody titer detection and specific pathogen PCR detection. Then, according to the pathogen results, adjust antibiotics
  Arms: Conventional pathogen detection
Drug: Meropenem，Imipenem，Caspofene，Osstat — Meropenem，Imipenem，Caspofene，Osstat

SUMMARY:
Investigators plan to conduct the participants level, 1:1 randomized trial at the Central ICU and respiratory ICU of Xiangya Hospital in Changsha, China, from January 1, 2018 to December 31, 2019. Participants with initial diagnosis of severe pneumonia will be first treated with empiric therapy, after 48-72 hours, the participants's condition will be evaluated, and participants who will have been initially cured and died should be excluded.The participants who will have failed the initial treatment will be then randomly divided into two groups: the NGS group and the conventional treatment group. Bronchoalveolar lavage fluid will be taken by bedside bronchoscopy when the participants underwent nasal high-flow oxygen therapy, non-invasive ventilation, and invasive ventilation,or venous blood will be taken for examination. Participants in the NGS group will be tested for both NGS and conventional pathogens, however, the routine group will be only routinely tested. According to the pathogen results, participants with non-severe pneumonia will be excluded, and medication should be adjusted under the joint guidance of infectious and respiratory specialists. Then investigators will compare the first outcome: 28-day mortality, and secondary outcome: ICU hospitalization time, mechanical ventilation time, Hospitalization costs, antibiotic use costs, SOFA scores, CURB-65 scores, APACHE scores, and other clinical indicators.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with severe pneumonia between the ages of 18 and 85 years; the diagnosis of severe pneumonia is based on IDSA / ATS

Exclusion Criteria:

* < 18 years old, received antibiotic treatment within 14 days before admission, suffering from severe immunosuppression, multi-drug resistance, refractory tuberculosis, end-stage renal disease or liver disease (uremia, advanced liver cancer), pregnancy. Besides, we need to rule out patients who have been improved, died, and abandoned during the initial treatment。

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
mortality | 28 day
  Using the Kaplan-Meier method to analyze the differences in mortality between the two groups within 28 days

SECONDARY OUTCOMES:
mechanical ventilation time | 30 days
  According to the secondary result, comprehensively evaluate the two detection methods for the treatment of patients with severe pneumonia

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China